CLINICAL TRIAL: NCT06348043
Title: Circulatory Support in Pediatric Heart Failure Patients Using the Jarvik 2015 LVAD: A Pivotal
Brief Title: Pumps for Kids, Infants and Neonates (PumpKIN): The Jarvik 2015 Pivotal Trial
Acronym: PumpKIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Texas (Other); Carelon Research (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Almond, Professor of Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU_PumpKIN; 1UG3HL163311-01A1 (NIH)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Pediatric HD, Stage IV; LVAD
Keywords: LVAD; Pediatric heart failure; advanced cardiac therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LVAD support with the Jarvik 2015 (Experimental): Children implanted with the Jarvik 2015 LVAD as a bridge to heart transplant
  Interventions: Device: Jarvik 2015 LVAD

INTERVENTIONS:
Device: Jarvik 2015 LVAD — Medical device used to treat children awaiting heart transplant who fail optimal medical therapy.

SUMMARY:
This is a 22-subject prospective, multicenter, single-arm clinical trial to evaluate the safety and effectiveness of the Jarvik 2015 left ventricular assist device (LVAD) as a bridge to heart transplant in children weighing 8 to 30 kilograms. Data generated from the study will be used to support FDA review and potential approval of the device under the Humanitarian Device Exemption (HDE) regulation, the FDA approval pathway for devices intended to treat rare and orphan diseases.

DETAILED DESCRIPTION:
This is a NHLBI-funded study is a prospective, multicenter, single-arm clinical trial to evaluate the safety and effectiveness of the Jarvik 2015 left ventricular assist device (LVAD) as a bridge to heart transplant in children where few LVAD options are available and require hospital confinement. Children weighing 8 to 30 kg will be eligible if they have end-stage heart failure refractory to medical therapy due to severe systolic dysfunction. Children with single ventricle heart disease, heart failure with preserved ejection fraction (HFpEF), those requiring BIVAD support, and those with irreversible end-organ dysfunction will be excluded. The primary probable benefit endpoint of the study is survival to heart transplant, recovery or 180 days of support in the absence of severe stroke. The primary safety endpoint of the study is freedom from any new symptomatic stroke. A total of 22 subjects will be enrolled in the trial at 14 sites in the US and Europe. Subjects will be enrolled over roughly 3 years (38 months) and followed for 1 year post explant. Data generated from the study will be used to support FDA review and potential approval of the device under the Humanitarian Device Exemption (HDE) regulation, the FDA approval pathway for devices intended to treat rare and orphan diseases. Children

ELIGIBILITY:
Inclusion Criteria:

Children with severe (Ross or New York Heart Association) class IV HF despite optimal medical therapy (Interagency Registry for Mechanically Assisted Circulatory Support [INTERMACS] profile 1 or 2 for pediatrics) who require mechanical circulatory support as a bridge to transplant and meet all the criteria below:

1. Males and females with body weight between 8 kg, and 30 kg
2. Body surface area (BSA) between 0.4 m2 and 1.0 m2
3. Two-ventricle circulation, including cardiomyopathy, repaired structural heart disease (e.g., anomalous left coronary artery from the pulmonary artery [ALCAPA], aortic stenosis) or acquired heart disease (e.g., , Kawasaki disease) 4. INTERMACS Profile 1 or 2 as evidenced by: a. Inability to wean from extra-corporeal membrane oxygenation (ECMO) or other temporary circulatory support (TCS), OR b.Inability to wean from mechanical ventilator support, OR c. Inotrope-dependent,decompensatedHFANDmeetoneormoreofthe following severity criteria within 48 hours prior to implant (unless otherwise noted), attributed to decompensated HF despite optimal medical therapy: i. Urine output <0.5 cc/kg/hour for 12hr ii. Creatinine level >2 times the upper limit of normal (ULN) for age iii. Alanine aminotransferase (ALT) or total bilirubin level >3 times the ULN for age (either qualifies the patient) iv. Mixed venous oxygen saturation (SvO2) <55% (or arteriovenous oxygen difference >45%) v. Acidosis: Base excess >-5 vi. Inability to tolerate appropriate enteral calories vii. Inability to ambulate or participate in age-appropriate activities of daily living (ADLs) and/or cardiac rehabilitation/physical therapy

5. LVAD support is intended for bridge-to transplant. Subject is listed for transplant or eligible (i.e., no medical or surgical contraindications) to be listed for cardiac transplant, United Network for Organ Sharing (UNOS) status 1A, or equivalent 6. Implant performed at a US or European site participating in the Jarvik 2015 IDE Pivotal Trial.

7. Written consent of parent(s) or legally authorized representative (LAR) where appropriate.

Exclusion Criteria:1. Severe right ventricular (RV) dysfunction or significant arrhythmia where treatment with a durable RV assist device (RVAD) (i.e., biventricular assist device) is definite or highly likely. 2. Complex cardiac anatomy including but not limited to:

1. Single ventricle anatomy
2. Presence of a mechanical heart valve
3. Unrepairable severe aortic insufficiency 3. Stable inotrope dependence (INTERMACS profile 3) 4. Severe or irreversible renal dysfunction, liver dysfunction or pulmonary dysfunction. 5. Known contraindication to systemic anticoagulation (e.g., coagulopathy) 6. CPR with duration >30 consecutive minutes within 48 hours prior to device implant or CPR with uncertain neurological status 7. ECMO use for >10 consecutive days 8. Known cerebrovascular event within the past 30 days or uncertain neurological status 9. Unmanageable bleeding per judgment of the investigator 10. Ventricular dysfunction that is likely to recover (e.g., acute myocarditis, metabolic myopathy where LV dysfunction is present solely with intermittent acidosis/crises).

   11. A non-dilated LV as determined by a left ventricular end-diastolic dimension or left ventricular end-diastolic volume z score of <+2.5 12. Systolic dysfunction that is not severe (LV ejection fraction of >35%) (e.g., heart failure with preserved ejection fraction, aka primary diastolic dysfunction). 12. Unresolved malignancy 13. Active, systemic infection unresponsive to antimicrobials therapy 14. Currently participating in an interventional trial whose protocol prevents effective application of the Jarvik 2015 device, potentially has an independent effect on trial endpoints, or otherwise interferes with execution of the PumpKIN protocol

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Survival to heart transplant, recovery or 180 days of support in the absence of severe stroke. | 180 days
  Patient survival to heart transplant, recovery or 180 days of support in the absence of severe stroke as defined by the Pediatric Stroke Outcomes Measure (PSOM, (range 0 to 10 with 0 no deficit to 10 maximum deficit) performed at 12 months post-explant. Severe stroke is defined an abnormal PSOM score due to stroke that meets the following criteria: PSOM score of 3-4 in Part A (sensory and motor assessment) OR Score of 3-4 in Parts B and C combined (language comprehension and language production) OR Score of 2 in Part D (cognitive or behavioral deficit).
Freedom from symptomatic stroke | 12 months post-explant
  Freedom from symptomatic stroke based on the 12-month Pediatric Stroke Outcome Measure (PSOM, symptomatic stroke defined as a PSOM >0 due to stroke, PSOM score range 0-10 with higher scores corresponding to more severe stroke injury). Participants meet criteria for no stroke if they do not meet ACTION criteria for stroke at 12 months or stroke is present with a PSOM score of 0).

SECONDARY OUTCOMES:
Incidence rate of all protocol-defined SAE's through 180 days of support definitely or probably related to the device | 180 days
  Incidence rate of all protocol-defined SAE's through 180 days of support definitely or probably related to the device using the ACTION definitions and rules for censoring and attribution, the industry standard in pediatric VAD therapy
Distribution of Pediatric Stroke Outcomes Measures | 12-months post explant for stroke occurring during the first 180 days of support
  Distribution of Pediatric Stroke Outcomes Measures (PSOM scores) in children with a new stroke diagnosis during the trial as assessed at 12 months post-explant.
The KOSCHI score | 12 months post-explant in children with strokes occurring during the first 180 days of support
  The Kings Outcomes Scale for Children Head Injury (KOSCHI) score (range 1-5, with 1-poor to 5-good functional state) for those diagnosed with a new stroke during the first 180 days as measured at 12 months post-explant.
Overall survival on Jarvik 2015 support to 180 days | 180 days
  Overall patient survival on Jarvik 2015 support without converting to a non-Jarvik device for left heart support (Kaplan-Meier estimate)

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Study Chair — Children's Healthcare of Atlanta

IPD SHARING:
Plan to Share IPD: No